CLINICAL TRIAL: NCT02938299
Title: A Pivotal Phase III, Open-label, Randomized, Controlled Multi-center Study of the Efficacy of L19IL2/L19TNF Neoadjuvant Intratumoral Treatment Followed by Surgery Versus Surgery Alone in Clinical Stage III B/C Melanoma Patients
Brief Title: Neoadjuvant L19IL2/L19TNF- Pivotal Study
Acronym: Pivotal
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2TNF-02/15
Record Dates: First submitted 2016-10-11; First posted 2016-10-19 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — daromun; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: neoadjuvant + surgery (Experimental): Patients in Arm 1 will receive multiple intratumoral administrations into all injectable cutaneous, subcutaneous, and nodal tumors of a mixture of L19IL2 and L19TNF once weekly for up to 4 weeks (or until all injectable tumors have disappeared, or intolerance to study treatment or in the opinion of the investigator immediate surgical resection or any other treatment for melanoma is warranted, whichever occurs first).
  Newly occurring injectable melanoma lesions within the 4 weeks treatment period will also be treated as described. Surgical resection of all existing metastases will follow within 4 weeks after end of treatment. Surgery will be performed after the safety evaluation carried out at week 5 and, if indicated, may be carried out on the same day of the safety evaluation.
  Interventions: Drug: L19IL2 + L19TNF; Procedure: Surgery
- Arm 2: surgery alone (Active Comparator): Patients in Arm 2 will receive directly surgical resection of melanoma tumor lesions within 4 weeks after randomization.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: L19IL2 + L19TNF — Mixture of L19IL2 and L19TNF once weekly
  Arms: Arm 1: neoadjuvant + surgery
Procedure: Surgery — Surgical resection of melanoma tumor lesions

SUMMARY:
Phase III, open-label, randomized, controlled multi-center study of the efficacy of L19IL2/L19TNF neoadjuvant intratumoral treatment in Stage III B/C melanoma patients.

DETAILED DESCRIPTION:
Phase III, open-label, randomized, controlled multi-center study. In the study, 214 patients will be enrolled and parallel assigned (via automated randomization system) in a 1:1 fashion to one of two different arms:

ARM 1:

Patients in Arm 1 will receive multiple intratumoral administrations into all injectable cutaneous, subcutaneous, and nodal tumors of a mixture of L19IL2 and L19TNF once weekly for up to 4 weeks (or until all injectable tumors have disappeared, or intolerance to study treatment or in the opinion of the investigator immediate surgical resection or any other treatment for melanoma is warranted, whichever occurs first). The whole volume of L19IL2/L19TNF will be distributed among all injectable lesions.

Newly occurring injectable melanoma lesions within the 4 weeks treatment period will also be treated as described. For the new lesions the treatment period will not be extended beyond the pre-defined 4 week- treatment period with a clock start at the time of the first intralesional L19IL2/L19TNF injection. Surgical resection of all existing metastases will follow within 4 weeks after end of treatment. Surgery will be performed after the safety evaluation carried out at week 5 and, if indicated, may be carried out on the same day of the safety evaluation.

Post-surgery EMA-approved adjuvant therapy is allowed at discretion of the treating physician.

ARM 2:

Patients in Arm 2 will receive directly surgical resection of melanoma tumor lesions within 4 weeks after randomization.

Post-surgery EMA-approved adjuvant therapy is allowed at discretion of the treating physician.

Patients will be followed on a regular basis for the primary outcome until 36 months from randomization and up to 60 months for overall survival.

Expected patient enrollment interval: 60 months. Duration of individual patient's participation: up to 60 months. End of treatment corresponds to the day of surgery for patients randomized to both Arm 1 and Arm 2.

End of study corresponds to the last patient last visit (LPLV). The final primary efficacy analysis will be conducted when the 95th recurrence event is observed.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of malignant melanoma of the skin with locally advanced disease as defined by clinical stage III B and III C according to AJCC 7th Ed., eligible for complete surgical resection.
2. Eligible subjects must have measurable disease and must be candidate for intralesional therapy with at least one injectable cutaneous, subcutaneous, or nodal melanoma lesion (≥ 10 mm in longest diameter) or with multiple injectable lesions that in aggregate have a longest diameter of ≥ 10 mm.
3. Prior anti-tumor treatment for the primary melanoma lesion, including surgery and approved adjuvant treatments (e.g., radiotherapy, immune checkpoint inhibitors, BRAF/MEK inhibitors, etc.) is allowed.
4. Males or females, age ≥ 18 years.
5. ECOG Performance Status/WHO Performance Status ≤ 1.
6. Life expectancy of at least 24 months (see paragraph 6.3.1).
7. Absolute neutrophil count > 1.5 x 109/L.
8. Hemoglobin > 9.0 g/dL.
9. Platelets > 100 x 109/L.
10. Total bilirubin ≤ 30 µmol/L (or ≤ 2.0 mg/dl).
11. ALT and AST ≤ 2.5 x the upper limit of normal (ULN).
12. Serum creatinine < 1.5 x ULN.
13. LDH serum level ≤ 1.5 x ULN.
14. Documented negative test for HIV, HBV and HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV (e.g., anti-HBsAg and/or anti-HBc Ab) negative serum HBV-DNA is also required.
15. All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) Grade ≤ 1 unless otherwise specified above.
16. Negative pregnancy test at screening for Women Of Childbearing Potential (WOCBP*). Pregnant women are not allowed to participate to this study. WOCBP must be using, from the screening to three months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Pregnancy test will be repeated at the Safety Visit (only WOCBP and only for patients in Arm 1).
17. Male patients with WOCBP partners must agree to use simultaneously two acceptable methods of contraception (i.e., spermicidal gel plus condom) from the screening to three months following the last study drug administration.
18. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
19. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion Criteria:

1. Uveal melanoma, mucosal melanoma or melanoma with unknown primary.
2. Evidence of distant metastases at screening.
3. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1), second primary melanoma in situ or any cancer curatively treated ≥ 5 years prior to study entry.
4. Presence of active infections (e.g., requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
5. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
6. Inadequately controlled cardiac arrhythmias including atrial fibrillation.
7. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
8. LVEF ≤ 50% and/or abnormalities observed during baseline ECG and Echocardiogram investigations that are considered as clinically significant by the investigator.
9. Uncontrolled hypertension.
10. Ischemic peripheral vascular disease (Grade IIb-IV).
11. Severe diabetic retinopathy.
12. Active autoimmune disease.
13. History of organ allograft or stem cell transplantation.
14. Recovery from major trauma including surgery within 4 weeks prior to enrollment.
15. Known history of allergy to IL2, TNF, or other human proteins/peptides/antibodies or any other constituent of the product.
16. Breast feeding female.
17. Anti-tumor therapy (except allowed treatments listed at point 3 of Inclusion criteria) within 4 weeks before enrollment.
18. Previous in vivo exposure to monoclonal antibodies for biological therapy (except allowed treatments listed at point 3 of Inclusion criteria) in the 6 weeks before enrollment.
19. Planned administration of growth factors or immunomodulatory agents (except allowed treatments listed at point 3 of Inclusion criteria) within 7 days before enrollment.
20. Patient requiring or taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
21. Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.
22. Previous enrolment and randomization in this same study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) rate | 1 year after randomization
  Recurrence-free survival (RFS) in the treatment arm (L19IL2/L19TNF plus surgery; Arm 1) versus control arm (Arm 2).

SECONDARY OUTCOMES:
Local recurrence-free survival (LRFS) | 1year, 2years, 3years after randomization and 1year after surgery
Distant metastasis-free survival (DMFS) rate | 1year, 2years, 3years after randomization and 1year after surgery
Recurrence-free survival (RFS) rate | 2years, 3years after randomization
Overall survival (OS) | 1year, 2years, 3years after randomization
Percentage of Participants With On-Study Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 3 years
Percentage of Participants With Worst On-Study Hematological and Chemistry Abnormalities | up to 36 months
Clinically Meaningful Changes in Vital Signs and Physical Examinations | up to 36 months
Changes in absolute counts and relative percentages of lymphocytic subpopulations over time | (1) At screening, (2) At Day of surgery: from Day 1 to Day 54, (3) After 3 months from surgery: Day 91 to Day 144
  Immunophenotypic characterization of PBMCs for changes in absolute counts and relative percentages of lymphocytic subpopulations (e.g., Tregs, MDSCs etc.) over time (only for patients recruited in German centers).
HAFA | (1) At Day 1, (2) At Day 29, (3) After 3 months from surgery: Day 119 to Day 144
  Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19IL2 and L19TNF.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina C. Kähler, MD, Principal Investigator — University Hospital Schleswig-Holstein; Mario Santinami, MD, Principal Investigator — Istituto Nazionale Tumori Milano; Piotr Rutkowski, MD, Principal Investigator — Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie Warszawa; Caroline Robert, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (22):
- France (3):
  - Hôpital de la Timone, Marseille
  - Hôpital Universitaire de Nantes, Nantes
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Dresden
  - Hauttumorzentrum Hannover (HTZH), Hanover, Hannover
  - Heidelberg University Hospital, Heidelberg, Heidelberg
  - Kiel University Hospital, Kiel, Kiel
  - Leipzig University Hospital, Leipzig, Leipzig
  - Charité Campus Mitte (CCM), Berlin, State of Berlin
  - Tübingen University Hospital, Tübingen, Tübingen
  - Klinik für Dermatologie und Allergologie, Universitätsklinikum Augsburg, Augsburg
  - Klinik für Dermatologie, Medizinische Fakultät Universitätsklinikum Essen, Essen
  - Klinik und Polyklinik für Dermatologie, Universitätsklinikum Regensburg, Regensburg
- Italy (7):
  - IRCCS A.O.U. San Martino - IST, Genova, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan
  - Istituto Oncologico Veneto, IRCCS, Padua, Padova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Naples
  - AOU Senese, Siena
  - ASUGI Trieste, Trieste
  - AOU Città della Salute e della Scienza, Turin
- Poland (2):
  - Medgart Centrum Medyczne, Gdansk
  - Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie Warszawa, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahler KC, Hassel JC, Ziemer M, Rutkowski P, Meier F, Flatz L, Gaudy-Marqueste C, Zimmer L, Santinami M, Russano F, von Wasielewski I, Eigentler TK, Maio M, Zalaudek I, Haferkamp S, Quaglino P, Welzel J, Rocken C, Enk A, Simon JC, Switaj T, Garzarolli M, Amaral T, Malissen N, Livingstone E, Elia G, Covelli A, Lorizzo K, Neri D, Mulatto S, Parca A, Pizzichi B, Ascierto PA, Garbe C, Robert C, Schadendorf D, Hauschild A. Neoadjuvant intralesional targeted immunocytokines (daromun) in stage III melanoma. Ann Oncol. 2025 Oct;36(10):1166-1177. doi: 10.1016/j.annonc.2025.06.014. Epub 2025 Jul 7. PMID 40633690
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215